CLINICAL TRIAL: NCT05288348
Title: DSUVIA Early Evaluation of PAIN (DEEP) Trial
Brief Title: DSUVIA Early Evaluation of Pain Trial
Acronym: DEEP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Frank Guyette (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Frank Guyette, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY21100180; W81XWH-16-D-0024 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2022-02-22; First posted 2022-03-21 (Actual); Results first posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Traumatic Injury
MeSH Terms: conditions — Wounds and Injuries | interventions — Sufentanil; Administration, Sublingual

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- DSUVIA (sufentanil) (Experimental): Subjects will receive a single dose of 30 micrograms DSUVIA (sufentanil) tablet utilizing a sublingual applicator
  Interventions: Drug: Sufentanil 30 MCG Sublingual Tablet
- Standard Care (Active Comparator): Subjects will receive standard care pain management
  Interventions: Drug: standard care pain treatment

INTERVENTIONS:
Drug: Sufentanil 30 MCG Sublingual Tablet — 30 microgram sublingual tablet administered using sublingual applicator
  Arms: DSUVIA (sufentanil)
Drug: standard care pain treatment — standard care pain treatment given in Emergency Department
  Arms: Standard Care

SUMMARY:
Randomized, interventional trial of Emergency Department (ED) administration of DSUVIA (sufentanil) versus standard care pain management comparing pain treatment outcomes in injured patients with moderate to severe pain

ELIGIBILITY:
Inclusion Criteria:

1. Trauma activation (Level I, II or III)
2. Age 18-70 years inclusive
3. Need for pain treatment based upon NRS (0-100) clinical pain measurement ≥ 50
4. Estimated time in Emergency Department > 30 minutes following informed consent

Exclusion Criteria:

1. Advanced airway management prior to 1st dose administration
2. Known allergy to opioids
3. Known prisoner
4. Known pregnancy
5. ED pain medication contraindicated
6. Significant respiratory depression
7. Known or suspected gastrointestinal obstruction, including paralytic ileus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2024-01-21 (Actual); Study Completion 2024-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Sperry, MD, Study Director — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with the funding agency as well as other researchers upon request to the Principal Investigator
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available after publication of the primary manuscript
Access Criteria: Requests for data will be submitted in writing and reviewed by the principal Investigator

REFERENCES:
- [Derived] Guyette FX, Chaudhary P, Vincent LE, Love ET, Brubaker DP, Neal MD, Brown JB, Rixe J, Barton DJ, Yates A, Wisniewski SR, Sperry JL. A Randomized Controlled Trial of Sublingual Sufentanil in Early Management of Pain in Trauma. Anesth Analg. 2025 Jul 1;141(1):172-180. doi: 10.1213/ANE.0000000000007384. Epub 2025 Feb 7. PMID 39919020

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DSUVIA (Sufentanil) | Standard Care
Started | 76 | 74
Completed | 76 | 74
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DSUVIA (Sufentanil) | Standard Care | Total
Number analyzed (Participants) | 76 | 74 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (16) | 48 (14) | 48 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 52 | 50 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 61 | 62 | 123
  Unknown or Not Reported | 14 | 11 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 16 | 21
  White | 64 | 55 | 119
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 3 | 10
Total Glascow Coma Scale [Mean (Standard Deviation); unit: units on a scale] — The scale is the Glasgow Coma Scale. The Total score (Range 3-15) is the sum of the Eye (Range 1-4) Verbal (Range 1-5) and Motor (Range 1-6) scores, higher numbers in the sub scale are better. GCS Total of 15 is the best outcome while GCS 3 is worst and unresponsive. All patients enrolled in the study had to be capable of informed consent and therefore all had a GCS of 15.
  units on a scale | 15 (0) | 15 (0) | 15 (0)
Injury Severity Score [Median (Inter-Quartile Range); unit: units on a scale] — The scale is the Injury Severity Score. The Total ISS score (Range 0-75) is the sum of the squares of the three worst Abbreviated Injury Scores (AIS) from six body regions: Head/Neck (Range 0-5) Face (Range 0-5) Chest (Range 0-5), Abdomen (Range 0-5), Extremity (Range 0-5) and External (Range 1-5) scores, higher numbers in the sub scale are associated with worse injury. An AIS score of 0 indicates no injury, a score of 5 indicates a critical injury. The ISS Total is associated with mortality risk.
  units on a scale | 5 [4 to 9] | 5.5 [4 to 9] | 5 [4 to 9]
Injury Type [Count of Participants; unit: Participants]
  Blunt | 73 | 71 | 144
  Penetrating | 3 | 2 | 5
  Both | 0 | 1 | 1
Verbal Numerical Rating Scale @ 0 min [Mean (Standard Deviation); unit: units on a scale] — The scale Verbal Numerical Rating Scale (VNRS). The VNRS score (Range 0-100) is the patients assessment of their pain on a scale of 0 (no pain) to 100 (the most pain imaginable).
  units on a scale | 81 (15) | 81 (14) | 81 (15)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 136 (20) | 136 (23) | 136 (21)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 79 (23) | 86 (18) | 83 (21)
Heart Rate [Mean (Standard Deviation); unit: beats per minute] | 82 (15) | 83 (15) | 83 (15)

OUTCOME MEASURES:

1. Primary Outcome: Verbally Administered Numeric Rating Scale (VNRS)
Description: Verbally administered Numeric Rating Scale (VNRS) for clinical pain measurement (scale of 0-100, where 0 is having no pain)
Time Frame: 30 minutes after administration
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DSUVIA (Sufentanil) | Standard Care
Number analyzed (Participants) | 76 | 74
units on a scale | 68 (27) | 66 (23)
Statistical Analysis 1: Comparison: DSUVIA (Sufentanil) vs Standard Care; Test type: Superiority; p = 0.56, Mixed Models Analysis — unadjusted; Mixed methods ANOVA; Mean Difference (Final Values) = 2.57, 95% CI 2-sided [-6.19 to 11.33]
Statistical Analysis 2: Comparison: DSUVIA (Sufentanil) vs Standard Care; Adjusted for age, sex, respiratory rate and injury type; Test type: Superiority; p = 0.92, Mixed Models Analysis; Mixed methods ANOVA; Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-10.5 to 9.48]

2. Secondary Outcome: Verbally Administered Numeric Rating Scale (VNRS)
Description: as for outcome 1
Time Frame: Every 30 min from 30 min post administration until the time of ED discharge or rescue narcotic administered and up to 120 minutes after administration, whichever comes first
Population: The number of patients analyzed at subsequent time points decreases as patients received rescue medications or left the Emergency Department (for admission, operative intervention, or discharge) prior to the 2 hr follow up period.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DSUVIA (Sufentanil) | Standard Care
Number analyzed (Participants) | 76 | 74
units on a scale
  30 minutes | 68 (27) | 66 (23)
  60 minutes: number analyzed (Participants) | 52 | 50
  60 minutes | 59 (29) | 66 (27)
  90 minutes: number analyzed (Participants) | 40 | 37
  90 minutes | 53 (29) | 64 (27)
  120 minutes: number analyzed (Participants) | 36 | 27
  120 minutes | 53 (30) | 62 (28)
Statistical Analysis 1: Comparison: DSUVIA (Sufentanil) vs Standard Care; VNRS @ 60min; Test type: Superiority; p = 0.18, Mixed Models Analysis; Mixed effects ANOVA; Mean Difference (Final Values) = -7.14, 95% CI 2-sided [-17.66 to 3.37]
Statistical Analysis 2: Comparison: DSUVIA (Sufentanil) vs Standard Care; VNRS @ 60 min Adjusted for sex and injury type; Test type: Superiority; p = 0.63, Mixed Models Analysis; Mixed effects ANOVA; Median Difference (Final Values) = 2.92, 95% CI 2-sided [-9.30 to 15.10]
Statistical Analysis 3: Comparison: DSUVIA (Sufentanil) vs Standard Care; VNRS @ 90 min; Test type: Superiority; p = 0.08, Mixed Models Analysis — Unadjusted; Mean Difference (Final Values) = -10.59, 95% CI 2-sided [-22.39 to 1.21]
Statistical Analysis 4: Comparison: DSUVIA (Sufentanil) vs Standard Care; VNRS @90min adjusted; Test type: Superiority; p = 0.28, Mixed Models Analysis; Mixed Method ANOVA; Mean Difference (Final Values) = 7.36, 95% CI 2-sided [-6.13 to 20.80] — Adjusted for ISS
Statistical Analysis 5: Comparison: DSUVIA (Sufentanil) vs Standard Care; VNRS @ 120 min; Test type: Superiority; p = 0.18, Mixed Models Analysis; Mean Difference (Final Values) = -9.52, 95% CI 2-sided [-23.60 to 4.56]
Statistical Analysis 6: Comparison: DSUVIA (Sufentanil) vs Standard Care; VNRS @ 120min adjusted for sex, HR, RR, and injury type; Test type: Superiority; p = 0.50, Mixed Models Analysis; Mixed Method ANOVA; Mean Difference (Final Values) = -5.24, 95% CI 2-sided [-20.70 to 10.20]

3. Secondary Outcome: Patient Global Assessment (PGA) of Pain Control
Description: An assessment of the patient's pain, made by the patient themselves, made at 30 minute intervals up to 120 min after the intervention, or until discharge, or administration of rescue medication
Time Frame: every 30 minutes after administration until the time of ED discharge or rescue narcotic administered, whichever comes first (up to 120 minutes after administration)
Population: Patient Global Assessment of Pain Control at 30 min
Measure: Count of Participants; unit: Participants
Arm/Group | DSUVIA (Sufentanil) | Standard Care
Number analyzed (Participants) | 66 | 63
Participants
  30 min: Poor | 22 | 12
  30 min: Fair | 21 | 14
  30 min: Good | 17 | 24
  30 min: Excellent | 6 | 13
  60 min: number analyzed (Participants) | 52 | 50
  60 min: Poor | 14 | 11
  60 min: Fair | 15 | 14
  60 min: Good | 15 | 14
  60 min: Excellent | 8 | 11
  90 min: number analyzed (Participants) | 40 | 37
  90 min: Poor | 8 | 6
  90 min: Fair | 12 | 11
  90 min: Good | 12 | 14
  90 min: Excellent | 8 | 6
  120 min: number analyzed (Participants) | 36 | 27
  120 min: Poor | 6 | 5
  120 min: Fair | 13 | 7
  120 min: Good | 9 | 8
  120 min: Excellent | 8 | 7
Statistical Analysis 1: Comparison: DSUVIA (Sufentanil) vs Standard Care; Test type: Superiority; p = 0.005, Chi-squared — PGA @ 30 min

4. Secondary Outcome: Time-weighted Summed Pain Intensity Difference (SPID) @ 30, 60, 90, 120 Min
Description: time-weighted Summed Pain Intensity Difference (SPID) is a statistical measure that calculates the cumulative pain reduction over a period of time by summing up the differences between baseline pain and current pain at various time points. The range for the SPID is 0-100 per time point, A score of 0 indicates no pain, a score of 100 indicating the worst pain intensity difference. Some patients did not participate in the SPID due to discharge or requiring rescue narcotic administration.
Time Frame: every 30 minutes after administration until ED discharge or rescue narcotic administered, whichever comes first (up to 120 minutes after administration)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DSUVIA (Sufentanil) | Standard Care
Number analyzed (Participants) | 69 | 72
units on a scale
  30 min | 6 (10) | 7 (10)
  60 min | 14 (20) | 14 (20)
  90 min | 22 (31) | 22 (30)
  120 min | 30 (42) | 30 (42)
Statistical Analysis 1: Comparison: DSUVIA (Sufentanil) vs Standard Care; SPID 30 last observation carried forward (LOCF) imputation technique to fill out the missing values by carrying forward the last observed value; Test type: Superiority; p = 0.39, General Addative Model; Odds Ratio (OR) = 1.45, 95% CI 2-sided [-4.77 to 1.89]
Statistical Analysis 2: Comparison: DSUVIA (Sufentanil) vs Standard Care; SPID 30, Adjusted Analysis last observation carried forward (LOCF) imputation technique to fill out the missing values by carrying forward the last observed value; Test type: Superiority; p = 0.29, General Additive Model; Odds Ratio (OR) = 1.72, 95% CI 2-sided [-1.50 to 4.95]
Statistical Analysis 3: Comparison: DSUVIA (Sufentanil) vs Standard Care; SPID @ 60min last observation carried forward (LOCF) imputation technique to fill out the missing values by carrying forward the last observed value; Test type: Superiority; p = 0.98, Generalized Additive Model; Odds Ratio (OR) = 0.08, 95% CI 2-sided [-6.63 to 6.47]
Statistical Analysis 4: Comparison: DSUVIA (Sufentanil) vs Standard Care; SPID 60 Adjusted Last observed carried forward to address missingness; Test type: Superiority; p = 0.85, Generalized Additive Model; Odds Ratio (OR) = 0.61, 95% CI 2-sided [-5.76 to 6.98]
Statistical Analysis 5: Comparison: DSUVIA (Sufentanil) vs Standard Care; SPID @ 90 mn last observation carried forward (LOCF) imputation technique to fill out the missing values by carrying forward the last observed value; Test type: Superiority; p = 0.8, Generalized Additive Model; Odds Ratio (OR) = -1.26, 95% CI 2-sided [-8.75 to 11.28]
Statistical Analysis 6: Comparison: DSUVIA (Sufentanil) vs Standard Care; SPID 90 min Adjusted last observation carried forward (LOCF) imputation technique to fill out the missing values by carrying forward the last observed value; Test type: Superiority; p = 0.92, Generalized Additive Model; Odds Ratio (OR) = -0.44, 95% CI 2-sided [-10.2 to 9.92]
Statistical Analysis 7: Comparison: DSUVIA (Sufentanil) vs Standard Care; SPID @ 120 min last observation carried forward (LOCF) imputation technique to fill out the missing values by carrying forward the last observed value; Test type: Superiority; p = 0.64, Generalized Additive Model; Odds Ratio (OR) = -3.18, 95% CI 2-sided [-10.45 to 16.90]
Statistical Analysis 8: Comparison: DSUVIA (Sufentanil) vs Standard Care; SPID 120 Adjusted last observation carried forward (LOCF) imputation technique to fill out the missing values by carrying forward the last observed value; Test type: Superiority; p = 0.75, Generalized Additive Model; Odds Ratio (OR) = -2.15, 95% CI 2-sided [-15.60 to 11.30]

5. Secondary Outcome: Number of Participants Who Needed Rescue Narcotic Doses
Description: Count of patients requiring additional pain medication after recieving the intervention (sufentanil) or the standard care control.
Time Frame: at 30 minutes following administration and during ED stay (up to 120 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | DSUVIA (Sufentanil) | Standard Care
Number analyzed (Participants) | 76 | 74
Participants | 27 | 29
Statistical Analysis 1: Comparison: DSUVIA (Sufentanil) vs Standard Care; Test type: Superiority; p = 0.64, two sided test of proportion; z statistic = 0.46, 95% CI 2-sided [-1.96 to 1.96]

6. Secondary Outcome: Patient Cognitive Function as Assessed by Six Item Screener (SIS)
Description: The Six Item Screener (SIS) is a simple assessment of cognitive impairment. It asks 6 questions, 3 based on recall and 3 based on orientation, each question is worth 1 point. The score can range between 0 and 6 correct answers. Higher numbers of correct answers indicated better outcomes (less cognitive impairment). Fewer patients were able to complete the SIS questionnaire then were enrolled in the study as some were discharged, received rescue medication or declined to participate prior to administration of the survey.
Time Frame: at 30 minutes following administration
Measure: Count of Participants; unit: Participants
Arm/Group | DSUVIA (Sufentanil) | Standard Care
Number analyzed (Participants) | 66 | 63
Participants
  6 Correct | 20 | 22
  5 Correct | 7 | 8
  4 Correct | 5 | 4
  3 Correct | 4 | 4
  2 Correct | 4 | 3
  1 Correct | 8 | 2
  0 Correct | 18 | 20
Statistical Analysis 1: Comparison: DSUVIA (Sufentanil) vs Standard Care; Test type: Superiority; p = 0.61, General Additive Models; Odds Ratio (OR) = -0.22, 95% CI 2-sided [-1.11 to 0.66]
Statistical Analysis 2: Comparison: DSUVIA (Sufentanil) vs Standard Care; 6 item screener adjusted analysis; Test type: Superiority; p = 0.54, General Additive Model; Odds Ratio (OR) = -0.28, 95% CI 2-sided [-1.23 to 0.65]

7. Secondary Outcome: Healthcare Professional Global Assessment (HPGA) of Method of Pain Control
Description: Acceptability of pain treatment to health care providers based on a subjective assessment of the patients facial expressions, behavior, physical presentation and reported pain level. Nurses caring for the participant following treatment with the study drug were asked to characterize their patients pain relief as Poor, Fair, Good or Excellent.
Time Frame: at 30 minutes following administration
Measure: Count of Participants; unit: Participants
Arm/Group | DSUVIA (Sufentanil) | Standard Care
Number analyzed (Participants) | 66 | 64
Participants
  Poor | 14 | 5
  Fair | 19 | 14
  Good | 23 | 28
  Excellent | 10 | 17
Statistical Analysis 1: Comparison: DSUVIA (Sufentanil) vs Standard Care; Healthcare Professional Global Assessment of method of pain control at 30 min; Test type: Superiority; p = 0.009, Ordinal Polytomous Logisitic Regression; Odds Ratio (OR) = 2.35, 95% CI 2-sided [1.24 to 4.46]
Statistical Analysis 2: Comparison: DSUVIA (Sufentanil) vs Standard Care; Healthcare Professional Global Assessment of method of pain control at 30 min. adjusted for ISS and Race; Test type: Superiority; p = 0.01, Ordinal polytomous logistic regression; Odds Ratio (OR) = 2.24, 95% CI 2-sided [1.18 to 4.29]

8. Secondary Outcome: Number of Participants With Hypoxia Needing Supplemental Oxygen
Description: The number of patients with an SpO2 less than 90 percent receiving supplemental oxygen
Time Frame: from administration to ED discharge or rescue narcotic administered, whichever comes first (up to 120 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | DSUVIA (Sufentanil) | Standard Care
Number analyzed (Participants) | 76 | 74
Participants | 4 | 4
Statistical Analysis 1: Comparison: DSUVIA (Sufentanil) vs Standard Care; Test type: Superiority; p = 0.96, Regression, Logistic; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.22 to 4.26]
Statistical Analysis 2: Comparison: DSUVIA (Sufentanil) vs Standard Care; Test type: Superiority; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.17 to 5.04] — Adjusted for age, sex and SpO2

9. Secondary Outcome: Number of Participants With Hypotension
Description: systolic blood pressure less than 90mmHg
Time Frame: from administration to ED discharge or rescue narcotic administered, whichever comes first (up to 120 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | DSUVIA (Sufentanil) | Standard Care
Number analyzed (Participants) | 76 | 74
Participants | 1 | 1
Statistical Analysis 1: Comparison: DSUVIA (Sufentanil) vs Standard Care; Test type: Superiority; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.04 to 24.92]
Statistical Analysis 2: Comparison: DSUVIA (Sufentanil) vs Standard Care; Test type: Superiority; Odds Ratio (OR) = 0.2, 95% CI 2-sided [0 to 14.28] — Adjusted for Heart Rate and Injury Severity Score

10. Secondary Outcome: Number of Participants With Nausea
Time Frame: from administration to ED discharge or rescue narcotic administered, whichever comes first (up to 120 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | DSUVIA (Sufentanil) | Standard Care
Number analyzed (Participants) | 76 | 74
Participants | 5 | 3
Statistical Analysis 1: Comparison: DSUVIA (Sufentanil) vs Standard Care; Test type: Superiority; Odds Ratio (OR) = 1.67, 95% CI 2-sided [0.39 to 8.37]
Statistical Analysis 2: Comparison: DSUVIA (Sufentanil) vs Standard Care; Test type: Superiority; Odds Ratio (OR) = 1.68, 95% CI 2-sided [0.39 to 8.60] — Adjusted for SpO2

11. Secondary Outcome: Number of Participants With Vomiting
Time Frame: from administration to ED discharge or rescue narcotic administered, whichever comes first (up to 120 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | DSUVIA (Sufentanil) | Standard Care
Number analyzed (Participants) | 76 | 74
Participants | 3 | 0

12. Secondary Outcome: Number of Participants With Headache
Time Frame: from administration to ED discharge or rescue narcotic administered, whichever comes first (up to 120 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | DSUVIA (Sufentanil) | Standard Care
Number analyzed (Participants) | 76 | 74
Participants | 1 | 2
Statistical Analysis 1: Comparison: DSUVIA (Sufentanil) vs Standard Care; Test type: Superiority; Odds Ratio (OR) = 0.48, 95% CI 2-sided [0.02 to 5.12]
Statistical Analysis 2: Comparison: DSUVIA (Sufentanil) vs Standard Care; Test type: Superiority; Odds Ratio (OR) = 0.41, 95% CI 2-sided [0.02 to 4.56] — Adjusted for heart rate

13. Secondary Outcome: Number of Participants With Dizziness Requiring Treatment
Description: Dizziness requiring treatment
Time Frame: from administration to ED discharge or rescue narcotic administered, whichever comes first (up to 120 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | DSUVIA (Sufentanil) | Standard Care
Number analyzed (Participants) | 76 | 74
Participants | 0 | 1
Statistical Analysis 1: Comparison: DSUVIA (Sufentanil) vs Standard Care; Test type: Superiority; p > 0.99, Chi-squared; difference of proportion = 0.135

14. Secondary Outcome: Number of Participants Who Had a 10 Point Reduction in VNRS Score @30 Min Intervals to 120min
Description: The Number of participants that had a 10 point reduction in their VNRS @ 30min intervals to 120min
Time Frame: Time to a 10 point reduction in VNRS following administration of study drug. Participants were followed to 120 min or discharge in 30 min intervals
Measure: Count of Participants; unit: Participants
Arm/Group | DSUVIA (Sufentanil) | Standard Care
Number analyzed (Participants) | 76 | 74
Participants
  Participants with a 10 point reduction @ 30 min | 28 | 36
  Participants with a 10 point reduction @ 60 min | 41 | 41
  Participants with a 10 point reduction @ 90 min | 42 | 43
  Participants with a 10 point reduction @ 120 min | 42 | 43
Statistical Analysis 1: Comparison: DSUVIA (Sufentanil) vs Standard Care; Test type: Superiority; p = 0.90, Regression, Cox; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.69 to 1.61]
Statistical Analysis 2: Comparison: DSUVIA (Sufentanil) vs Standard Care; Adjusted for Race and ISS; Test type: Superiority; p = 0.48, Regression, Cox; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.75 to 1.81]

15. Secondary Outcome: Number of Participants With Need for Bag Valve Mask Ventilation or Advanced Airway Management
Description: Need for advanced airway or bag valve mask ventilation
Time Frame: From drug administration up to 120 min following administration
Measure: Count of Participants; unit: Participants
Arm/Group | DSUVIA (Sufentanil) | Standard Care
Number analyzed (Participants) | 76 | 74
Participants | 0 | 0

16. Secondary Outcome: Richmond Agitation-Sedation Scale (RASS)
Description: The Richmond Agitation-Sedation Scale is scored from a -5 (unresponsive) to +4 (combative) with 0 being alert and calm.
Time Frame: Assessed at 30 minutes after administration
Population: RASS @ 30 min
Measure: Count of Participants; unit: Participants
Arm/Group | DSUVIA (Sufentanil) | Standard Care
Number analyzed (Participants) | 65 | 64
Participants
  RASS 4 @ 30 min | 0 | 0
  RASS 3 @ 30 min | 0 | 0
  RASS 2 @ 30 min | 1 | 0
  RASS 1 @ 30 min | 7 | 7
  RASS 0 @ 30 min | 46 | 48
  RASS -1 @ 30 min | 9 | 8
  RASS -2 @ 30 min | 2 | 0
  RASS -3 @ 30 min | 0 | 1
  RASS -4 @ 30 min | 0 | 0
  RASS -5 @ 30 min | 0 | 0
Statistical Analysis 1: Comparison: DSUVIA (Sufentanil) vs Standard Care; Test type: Superiority; p = 0.99, Non parametric General Addative Model; Odds Ratio (OR) = 0.00, 95% CI 2-sided [-0.15 to 0.15]
Statistical Analysis 2: Comparison: DSUVIA (Sufentanil) vs Standard Care; Adjusted; Test type: Superiority; p = 0.96, Non Parametric General Additive Model; Odds Ratio (OR) = 0.01, 95% CI 2-sided [-0.16 to 0.15]

17. Secondary Outcome: Richmond Agitation-Sedation Scale (RASS) @ 60 Min
Description: The Richmond Agitation-Sedation Scale is scored from a -5 (unresponsive) to +4 (combative) with 0 being alert and calm. Fewer patients were able to complete the SIS questionnaire then were enrolled in the study as some were discharged, received rescue medication or declined to participate prior to administration of the survey.
Time Frame: RASS @ 60 min
Measure: Count of Participants; unit: Participants
Arm/Group | DSUVIA (Sufentanil) | Standard Care
Number analyzed (Participants) | 52 | 50
Participants
  RASS 4 | 0 | 0
  RASS 3 | 0 | 0
  RASS 2 | 1 | 1
  RASS 1 | 3 | 4
  RASS 0 | 40 | 34
  RASS -1 | 5 | 9
  RASS -2 | 2 | 0
  RASS -3 | 0 | 2
  RASS -4 | 1 | 0
  RASS -5 | 0 | 0
Statistical Analysis 1: Comparison: DSUVIA (Sufentanil) vs Standard Care; Test type: Superiority; p = 0.84, Non Parametric General Additive Model; Odds Ratio (OR) = 0.01, 95% CI 2-sided [-0.17 to 0.16]
Statistical Analysis 2: Comparison: DSUVIA (Sufentanil) vs Standard Care; Adjusted; Test type: Superiority; p = 0.84, Non Parametric Generalized Additive Mode; Odds Ratio (OR) = 0.02, 95% CI 2-sided [-0.19 to 0.16]

18. Secondary Outcome: Richmond Agitation-Sedation Scale (RASS) @ 90 Min
Description: The Richmond Agitation-Sedation Scale is scored from a -5 (unresponsive) to +4 (combative) with 0 being alert and calm.Fewer patients were able to complete the SIS questionnaire then were enrolled in the study as some were discharged, received rescue medication or declined to participate prior to administration of the survey.
Time Frame: RASS @ 90 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | DSUVIA (Sufentanil) | Standard Care
Number analyzed (Participants) | 40 | 37
Participants
  RASS 4 | 0 | 0
  RASS 3 | 0 | 1
  RASS 2 | 0 | 0
  RASS 1 | 2 | 4
  RASS 0 | 32 | 25
  RASS -1 | 4 | 6
  RASS -2 | 2 | 1
  RASS -3 | 0 | 0
  RASS -4 | 0 | 0
  RASS -5 | 0 | 0
Statistical Analysis 1: Comparison: DSUVIA (Sufentanil) vs Standard Care; Test type: Superiority; p = 0.81, Non Parametric Generalized Additive Mode; Odds Ratio (OR) = 0.02, 95% CI 2-sided [-0.17 to 0.22]
Statistical Analysis 2: Comparison: DSUVIA (Sufentanil) vs Standard Care; Adjusted; Test type: Superiority; p = 0.91, Non Parametric Generalized Additive Mode; Odds Ratio (OR) = 0.01, 95% CI 2-sided [-0.20 to 0.22]

19. Secondary Outcome: Richmond Agitation-Sedation Scale (RASS) @ 120 Min
Description: as for outcome 17
Time Frame: RASS @ 120 min
Measure: Count of Participants; unit: Participants
Arm/Group | DSUVIA (Sufentanil) | Standard Care
Number analyzed (Participants) | 36 | 27
Participants
  RASS 4 | 0 | 0
  RASS 3 | 0 | 0
  RASS 2 | 0 | 0
  RASS 1 | 2 | 1
  RASS 0 | 32 | 20
  RASS -1 | 2 | 6
  RASS -2 | 0 | 0
  RASS -3 | 0 | 0
  RASS -4 | 0 | 0
  RASS -5 | 0 | 0
Statistical Analysis 1: Comparison: DSUVIA (Sufentanil) vs Standard Care; Test type: Superiority; p = 0.74, Non Parametric Generalized Additive Mode; Odds Ratio (OR) = 0.03, 95% CI 2-sided [-0.25 to 0.18]
Statistical Analysis 2: Comparison: DSUVIA (Sufentanil) vs Standard Care; Adjusted; Test type: Superiority; p = 0.63, Non Parametric Generalized Additive Mode; Odds Ratio (OR) = 0.05, 95% CI 2-sided [-0.30 to 0.18]

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 120 minutes after administration of the study drug
Description: Adverse events included hypoxia (SpO2 <90%) requiring supplemental oxygen, hypotension (SBP<90mmHg), need for bag mask ventilation or placement of an advanced airway. Episodes of nausea, vomiting, headache or dizziness requiring treatment also counted as an adverse event. Research assistants in the ED could identify these through direct observation, by report from the care team, or from sub sequence review of the medical record.
Arm/Group | DSUVIA (Sufentanil) | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/74
Serious Adverse Events (participants affected / at risk) | 7/76 | 6/74
Other Adverse Events (participants affected / at risk) | 5/76 | 4/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DSUVIA (Sufentanil) (N=76) | Standard Care (N=74)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) — SpO2 <90% requiring treatment
Hypotension (General disorders) | 1 (1) | 1 (1) — Systolic Blood Pressure <90mmHg
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) — Nausea requiring treatment
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) — Vomiting requiring treatment
Headache (Nervous system disorders) | 0 (0) | 0 (0) — Headache requiring treatment
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) — Dizziness requiring treatment
Need for an advanced airway (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) — Need for Bag Valve Mask ventilation or placement of an advanced airway
Need for Supplemental Oxygen to maintain SpO2 >90% (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DSUVIA (Sufentanil) (N=76) | Standard Care (N=74)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) — SpO2<90
Hypotension (General disorders) | 0 (0) | 0 (0) — SBP<90 mmHg
Nausea (Gastrointestinal disorders) | 4 (4) | 2 (2) — Nausea requiring treatment
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) — Vomiting requiring treatment
Headache (Nervous system disorders) | 1 (1) | 2 (2) — Requiring Treatment
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) — Requiring treatment
Need for supplemental oxygen (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) — Need for Oxygen to maintain SpO2>90%

LIMITATIONS AND CAVEATS:
Our study is a first of its kind comparing sublingual sufentanil to standard care in trauma patients. The intervention could not be blinded which imparts bias. This study was conducted at two level 1 trauma centers in the city of Pittsburgh and while the population was typical of our region, it may not be broadly generalizable. We did not dictate the choice or dose of analgesic in the standard arm. There was missingness in the data and no primary outcome was recorded in 20 subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT05288348/Prot_SAP_001.pdf
  • Informed Consent Form (2023-12-18): https://cdn.clinicaltrials.gov/large-docs/48/NCT05288348/ICF_000.pdf